CLINICAL TRIAL: NCT06699017
Title: Evaluation of the Effects of Continuous Anterior Chest Compression on Ventilation/Perfusion Ratios and Hemodynamics in SDRA
Brief Title: Effect of Continuous Anterior Chest Compression on Ventilation/Perfusion Ratio and Hemodynamics
Acronym: HemodyCACC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP230065
Record Dates: First submitted 2023-02-28; First posted 2024-11-21 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ARDS; cardiac output; ventilation perfusion ratio
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: Patient with moderate to severe ARDS under sedation and curarization keep on going
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with moderate to severe ARDS under sedation andcontinuous curarization (Experimental): Patient with moderate to severe ARDS under sedation andcontinuous curarization
  Interventions: Other: Continuous anterior chest compression

INTERVENTIONS:
Other: Continuous anterior chest compression — CACC is performed manually and the pressure applied will be maintained between 60 and 80 cmH2O.

SUMMARY:
Intro:

The mortality of acute respiratory distress syndrome (ARDS) remains high (40%), and may be aggravated by ventilation-induced lung injury (VILI), the main mechanisms of which are:

1. Anterior region overdistension,
2. Atelectrauma in the posterior regions. Positive expiratory pressure (PEEP) adjusted on the ventilator during ARDS aims to recruit posterior pulmonary territories in order to limit atelectrauma but is accompanied by a concomitant risk of overdistension of anterior territories.

Recent data suggest that continuous anterior chest compression (CACC) could limit the overdistension of the anterior regions by decreasing the compliance of the anterior chest wall and thus the regional transpulmonary pressure, while promoting the redistribution of ventilation to the posterior territories.

The effects of CCAC on ventilation/perfusion ratios and hemodynamics are unknown.

Hypothesis/Objective :

The participants hypothesize that during ARDS, CCAC:

1. Improves ventilation/perfusion ratios by decreasing both anterior territory dead space effect and posterior territory shunt,
2. Induce an improvement in cardiac output by decreasing right ventricular afterload (decrease in capillary compression related to the overdistension of the anterior territories and decrease in hypoxic vasoconstriction of the condensed territories).

Objective:

Primary outcome :

To evaluate the effects of CCAC on ventilation/perfusion ratios during moderate to severe ARDS.

Secondary outcome :

To evaluate the effects of CCAC on hemodynamics : left heart morphology, systolic and diastolic function, cardiac output, right heart morphology, systolic function, pulmonary hypertension, volemia.

Method In patient with moderate to severe ARDS, CACC is performed manually and the pressure applied will be maintained between 60 and 80 cmH2O.

Electrical impedance tomography of ventilation and perfusion will be used for the measurement of the percentage of areas with normal VA/Q ratios, areas of shunt and areas of dead space effect.

Left heart morphology, systolic and diastolic function, cardiac output, right heart morphology, systolic function, pulmonary hypertension, volemia will be evaluated by using echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ARDS moderate to severe according to the Berlin criteria
* Patient receiving continuous sedation and curarization
* Free and informed consent from the patient or family member

Exclusion Criteria:

* Pregnancy
* Adult patient subject to a legal protection measure (tutor, curator, etc.)
* Patients with a pacemaker, automatic implantable cardioverter defibrillator,
* Contraindications to thoracic belt placement (e.g., thoracic or spinal cord trauma, recent thoracic surgery)
* Undrained pneumothorax, bronchopleural fistula
* Hemodynamic instability (i.e., use of intravenous fluids of more than 10 mL/kg or vasopressors 2 mg/h of norepinephrine or 0.5 mg/h of epinephrine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
percentage of areas with normal VA/Q ratios, areas of shunt and areas of dead space effect. | 28 days
  demonstration that CACC may improve VA/Q ratio by using electrical impedance tomography

SECONDARY OUTCOMES:
CACC may induce a modification in cardiac output by decreasing right ventricular afterload | 28 days
  measurement of cardiac output with echocardiography via : left ventricle outflow tract velocity time integral cm)
CACC may induce a modification in patient with right ventricular injury | 28 days
  RV/LV : right ventricle end-diastolic ratio, to LV end-diastolic diameter ratio, sLV eccentricity index : systolic left ventricle eccentricity index; ACP : Acute cor pulmonale
CACC may induce a modification in right systolic function | 28 days
  measurement of right systolic function paramaters : TAPSE (mm) , S' annular tricuspid wave (m/s), RVFAC (%)
CACC may induce a modification in left systolic function | 28 days
  LVEF : left ventricular ejection fraction
CACC may induce a modification in ventilation distribution | 28 days
  ventilation distribution antero-posterior and right/left, assessed by electrical impedance tomography
CACC may induce a modification in lung perfusion distribution | 28 days
  lung perfusion distribution antero-posterior and right/left assessed by electrical impedance tomography

CONTACTS AND LOCATIONS:
Locations (1):
- Henri Mondor hospital, Créteil, Creteil, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION